CLINICAL TRIAL: NCT03104738
Title: A Comparison of the Impact of Basal Insulin Dosing Strategies on Next-day Surgery Blood Glucose Control
Brief Title: Basal Insulin Strategies Before Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Barbara Rogers, MD, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013H0232
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Results first posted 2018-11-05 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Open-label randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50% reduction of basal insulin dose (No Intervention): This is the institutional standard of care. The evening before surgery, 20 subjects will reduce their basal insulin dose to 50%.
- 25% reduction of basal insulin dose (Experimental): The evening before surgery, 20 subjects will reduce their basal insulin dose to 25%.
  Interventions: Other: 25% reduction of basal insulin dose

INTERVENTIONS:
Other: 25% reduction of basal insulin dose — Subjects will be instructed to reduce their basal insulin dose to 75% instead of our institutional 50%.
  Subject must check their own blood sugar before reporting to the hospital for their surgery. If the value is less than 70 or subjects are having symptoms of hypoglycemia, subjects will be instructed to immediately ingest 4-8 oz of fruit juice (without pulp) and call their doctor or the hospital.
  Arms: 25% reduction of basal insulin dose

SUMMARY:
Many patients with Type 2 Diabetes Mellitus (T2DM) are currently being managed with Basal Insulin (BI). However, there is little evidence to support guidelines on dosing adjustments in the preoperative period. The Society for Ambulatory Anesthesia does not advise a reduction in the dose of BI preoperatively, unless there is a specific history of hypoglycemia. The Endocrine Society suggests a 50% reduction in BI dose the evening before surgery. The authors hypothesized that a 25% reduction in BI dose the evening before surgery will result in better perioperative blood glucose control compared with our institutional 50% decrease.

DETAILED DESCRIPTION:
A total of 40 subjects diagnosed with T2DM taking once-daily evening BI, scheduled to undergo elective surgery under general anesthesia will be consented and randomized in a 1:1 ratio to received either 50% or 25% reduction of their regular evening BI dose on the evening before surgery. Blood glucose levels (BGL) will be recorded perioperatively according to institutional guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have volunteered and consented to participation in the study during their outpatient preoperative anesthesia appointment.
* Type II Diabetics taking once-daily evening basal insulin (glargine or detemir)
* Patients that will undergo general anesthesia
* Patients who have been on basal insulin for ≥ 3months

Exclusion Criteria:

* Inability to read, comprehend, and sign informed consent
* Patients with Type I Diabetes
* Patients who take short-acting insulin boluses which make up greater than 20% of their total daily insulin dose
* Patients who have been on chronic steroids ≥ 5 mg/dl prednisone daily or equivalent for ≥ 1 month within the past 12 months
* Pregnant patients
* Patients on twice-daily dosing of basal insulin
* Patient who take basal insulin in the morning
* Patients with a history of severe hypoglycemia, defined as any event in the previous year requiring assistance of another person to actively administer carbohydrate, glucagons, or other resuscitative actions
* Patients that will undergo cardiac, transplant, or brain surgeries
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Rogers, MD, Principal Investigator — Ohio State University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 25% Reduction of Basal Insulin Dose: The evening before surgery, 20 subjects will reduce their basal insulin dose to 25%.
  25% reduction of basal insulin dose: Subjects will be instructed to reduce their basal insulin dose to 75% instead of our institutional 50%.
  Subject must check their own blood sugar before reporting to the hospital for their surgery. If the value is less than 70 or subjects are having symptoms of hypoglycemia, subjects will be instructed to immediately ingest 4-8 oz of fruit juice (without pulp) and call their doctor or the hospital.
Period: Overall Study
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (11.4) | 57.9 (11.4) | 59.2 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 16 | 19 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Kg] | 105.9 (30.5) | 110.0 (23.3) | 108.0 (26.9)
Height [Mean (Standard Deviation); unit: cm] | 172.1 (11.7) | 166.4 (10.1) | 169.3 (11.2)
BMI [Mean (Standard Deviation); unit: Kg/m2] | 35.8 (10.2) | 39.9 (8.7) | 37.8 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Pre-operative Fasting Blood Glucose, as Measured by Standardized Point of Care Capillary Blood Glucose (CBG) Device in the Pre-op Holding Area.
Description: Capillary blood glucose before surgery, considering a fasting period up to 8 hours prior fasting blood glucose
Time Frame: Hospital arrival - Anesthesia start time. The time period did not exceed 4 hours, considering that surgeries were scheduled to be morning cases.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Number analyzed (Participants) | 20 | 20
mg/dl | 144.0 (39.0) | 152.5 (44.8)

2. Secondary Outcome: Incidence of Preoperative Hypoglycemia
Description: Capillary blood glucose level <80 mg/dl
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Number analyzed (Participants) | 20 | 20
Participants | 1 | 1

3. Secondary Outcome: Incidence of Preoperative Hypoglycemia Requiring Ingestion of Juice Prior to Arrival to the Hospital
Description: Capillary blood glucose level <70 mg/dl
Time Frame: Basal insulin dose administration the evening before surgery - Hospital arrival the morning of the surgery. The time period did not exceed 12 hours, considering a fasting period up to 8 hours and a preoperative period up to 4 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

4. Secondary Outcome: Incidence of Preoperative Hyperglycemia
Description: Capillary blood glucose level >179 mg/dl
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Number analyzed (Participants) | 20 | 20
Participants | 5 | 5

5. Secondary Outcome: Incidence of Intraoperative Hyperglycemia
Description: Capillary or arterial/venous blood glucose level >179 mg/dl
Time Frame: Anesthesia start time - Anesthesia stop time. The time period did not exceed 10 hours, considering type of surgeries or procedures.
Population: Out of 20 subjects in the 50% reduction, intraoperative blood glucose level for was not measured on 1 subject; therefore, only 19 subjects were analyzed for this outcome.
  Out of 20 subjects in the 25% reduction, intraoperative blood glucose level for was not measured on 3 subject; therefore, only 17 subjects were analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Number analyzed (Participants) | 19 | 17
Participants | 7 | 6

6. Secondary Outcome: Incidence of Patients Requiring Initiation of Perioperative IV Insulin Drip
Time Frame: Hospital arrival - 24 hours postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

7. Secondary Outcome: Incidence of Hyperglycemia in the Post-anesthesia Care Unit (PACU) to 24 Hours Post-operatively
Description: Capillary or arterial/venous blood glucose level >179 mg/dl
Time Frame: Anesthesia stop time - 24 hours postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Number analyzed (Participants) | 20 | 20
Participants | 9 | 15

8. Secondary Outcome: Incidence of Symptomatic Hypoglycemia Requiring Treatment in the PACU to 24 Hours Post-operatively
Description: Capillary or arterial/venous blood glucose level <70 mg/dl
Time Frame: Anesthesia stop time - 24 hours postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Number analyzed (Participants) | 20 | 20
Participants | 1 | 0

9. Secondary Outcome: Incidence of Hypoglycemia in the PACU to 24 Hours Post-operatively
Description: Capillary or arterial/venous blood glucose level <80 mg/dl
Time Frame: Anesthesia stop time - 24 hours postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Number analyzed (Participants) | 20 | 20
Participants | 1 | 5

10. Secondary Outcome: Incidence of Surgical Delay or Cancellation Due to Hyperglycemia
Time Frame: Hospital arrival - Surgery start date/time. The time period did not exceed 4 hours, considering that surgeries were scheduled to be morning cases
Measure: Count of Participants; unit: Participants
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

11. Secondary Outcome: Mean 24-hour Glucose Postoperatively
Time Frame: Anesthesia stop time - 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Number analyzed (Participants) | 20 | 20
mg/dl | 158.5 (31.7) | 165.2 (28.1)

ADVERSE EVENTS:
Time Frame: Since subject hospital arrival for the scheduled surgery until postoperative hour 24.
Arm/Group | 50% Reduction of Basal Insulin Dose | 25% Reduction of Basal Insulin Dose
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Intraoperative measurement of blood glucose was missing on 4 subjects. This measurement is Standard of care at our institution, nevertheless,on shorter surgeries this measurement was not perform, leading to missing data on this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes